CLINICAL TRIAL: NCT05654389
Title: Effectiveness of a New Pathway of Referring a Patient With Early Myocardial Infarction From Peripheral Hospital to Cardiac Centre in Hail, Saudi Arabia: A Randomized Clustered Trial
Brief Title: Effectiveness of Teleconsultation in Referring a Patient With Early Myocardial Infarction From Peripheral Hospital to Cardiac Centre in Hail, Saudi Arabia
Acronym: Telehealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The New Model of Care, Hail Health Cluster (Other Government)
Collaborators: Health Holding Company, Hail Health Cluster, Saudi Arabia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Model of Care
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Telemedicine
Keywords: telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of teleconsultation using WhatsApp to refer patient with with myocardial infarction (Experimental): Application of teleconsultation using WhatsApp for a patient with myocardial infarction with a provisional diagnosis of myocardial infarction during referral from a district hospital to a cardiac centre.
  Interventions: Other: Application of teleconsultation for a patient with a provisional diagnosis of myocardial infarction at the district hospital
- Routine care and handling of a patient with mycardial infarction at peripheral hospital (No Intervention): Routine care and consultation received by a patient with a provisional diagnosis of myocardial infarction during referral from the district hospital to the cardiac centre

INTERVENTIONS:
Other: Application of teleconsultation for a patient with a provisional diagnosis of myocardial infarction at the district hospital — Using teleconsultation for a patient with a provisional diagnosis of myocardial infarction during referral from the district hospital to the cardiac centre
  Arms: Application of teleconsultation using WhatsApp to refer patient with with myocardial infarction

SUMMARY:
The goal of this pragmatic trial is to test the benefit of using a teleconsultation for referring a patient with a heart attack at an early stage from the suburban hospital to the heart centre. A teleconsultation with an expert cardiologist will be conducted by the physician at a suburban hospital. The main questions it aims to answer are:

To what extent does the use of a teleconsultation for a patient with a heart attack work well in lowering the proportion of deaths among patients with heart attacks who will be referred from suburban hospitals to the heart centre? To what extent does the use of a teleconsultation for a patient with a heart attack work well in raising the proportion of stable cases with heart attacks who will be referred from suburban hospitals to the heart centre? Participants will be asked to participate in a teleconsultation referral pathway from the suburban hospital to the heart centre.

Researchers will compare the change in the proportion of death rate and survivors or stable cases in the intervention versus the control group during referral from suburban hospital to heart centre.

Making use of telehealth and smart applications will positively improve the quality of the provided health service at suburban hospitals where there is a limited number of specialized doctors.

DETAILED DESCRIPTION:
The economic burden of myocardial infarction is the highest in Saudi Arabia. This burden is mainly due to the associated costs of medical interventions and the length of hospital stay.

It is advisable that the health system in Saudi Arabia deploy appropriate measures for the prevention and early detection of myocardial infarction among diabetic patients. Otherwise, the economic burden of cardiovascular diseases is expected to shoot up.

A practical approach for referring patients with Myocardial Infarction (MI) is the modified meta-plan methodology for refereeing a patient from primary care to a cardiology clinic. This approach is recommended as an additional practical pathway for a patient with cardiovascular disease in primary care.

A concentrated value assessment model (CVAM) for determining percutaneous coronary intervention (PCI) levels is suggested to predict MI using accumulated sessions of ECG observation.

Patients at high risk of future myocardial infarction could be identified by every optician at the eye clinic using retinal images and demographic data,

Research Questions:

To what extent does the use of a teleconsultation intervention is effective in reducing the proportion of deaths among patients with myocardial infarction who will be referred from peripheral hospital to the cardiac centre? To what extent does the use of teleconsultation is effective in increasing the proportion of stable cases with myocardial infarction who will be referred from the peripheral hospital to the cardiac centre?

General objective:

To estimate the effectiveness of using a teleconsultation for patients with myocardial infarction at peripheral hospitals in reducing the proportion of deaths and increasing the proportion of stable cases among referral cases.

Specific Objectives:

Aim 1: To compare the proportion of death among cases with myocardial infarction who will be referred from a peripheral hospital to the cardiac centre in the intervention versus the control group (routine care).

Aim 2: To compare the proportion of stable cases of myocardial infarction who will be referred from the peripheral hospital to the cardiac centre in the intervention versus the control group (routine care).

Aim 3: To compare the proportion of cases who developed co-morbidities such as heart failure in the intervention versus the control group (routine care).

Literature Review:

A positive protective effect of antidepressant use to protect against developing myocardial infarction as primary care intervention is evident.

Research Design and Methods:

This is a six months clustered randomized trial that will recruit patients with provisional a diagnosis of myocardial infarction at a governmental peripheral hospital in Hail city.

Participants (P):

The participants will be adults presented to the physician at the peripheral hospital with symptoms and signs of myocardial infarction. The participants are expected to be adults aged 18 years and above. Children and young adults will be excluded. The aim is to report eligible cases by the physician at the peripheral hospital upon satisfaction with the written criteria for early MI diagnosis. The reporting will continue for six months from the beginning of the trial. Cases in both intervention and control clusters will be notified and reported regularly.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 to 80 with provisional diagnose of MI

Exclusion Criteria:

* severely ill patient and patient with other chronic conditions or cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of death among patients with myocardial infarction who will be referred from the peripheral hospital to the cardiac centre | 6 month from the start of the study
  The proportion of death among patients with myocardial infarction who will be referred from the peripheral hospital to the cardiac centre in the intervention versus the control group (routine care).
The proportion of stable cases of myocardial infarction who will be referred from the peripheral hospital to the cardiac centre | 6 month from the start of the study
  The proportion of stable cases of myocardial infarction who will be referred from the peripheral hospital to the cardiac centre in the intervention versus the control group (routine care).

SECONDARY OUTCOMES:
The proportion of stable cases of myocardial infarction who received Tissue Plasminogen Activator (TBA) before referral | 6 months after the start of the study
  The proportion of stable cases of myocardial infarction who received Tissue Plasminogen Activator (TBA) before referral from the peripheral hospital to the cardiac centre in the intervention group versus the control group (routine care).
The proportion of stable cases of myocardial infarction who developed co-morbidities | 6 months after the start of the study
  The proportion of stable cases of myocardial infarction who developed co-morbidities such as heart failure in the intervention versus the control group (routine care).

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Alshammari, VIP Chief MO, Study Chair — Hail Health Cluster; Fakhralddin Elfakki, Researcher at MOC, Principal Investigator — New Model of Care, Hail Health Cluser; Meshari Aljamani, MOC Lead, Study Director — New Model of Care, Hail Health Cluster

IPD SHARING:
Plan to Share IPD: No